CLINICAL TRIAL: NCT00889824
Title: Head-Mounted Vibrotactile Prosthesis for Patients With Chronic Postural Instability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barron Associates, Inc. (Industry); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0600; 1R43DC010080-01 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Dizziness
Keywords: Chronic imbalance; vestibular disorders; balance prosthesis
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prosthesis group (Experimental): balance prosthesis
  Interventions: Device: balance prosthesis

INTERVENTIONS:
Device: balance prosthesis — vibrotactile stimulation

SUMMARY:
The goal of this project is to provide individuals that have a balance deficit with a device that will give them signals that they can feel (vibrations) in order to help them maintain a correct sense of balance and perception of place in the environment.

DETAILED DESCRIPTION:
This proposal addresses a National Institute on Deafness and Other communication Disorders (NIDCD) research topic that emphasizes the "development of assistive devices for balance disorders". The proposed work will evaluate the assistive efficacy of such a balance prosthesis in a population of chronic imbalance patients spanning a wide range of disease etiologies.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients who have had chronic imbalance for at least one year, and have reached a functional performance plateau with respect to their balance adaptation.

Exclusion Criteria:

* Neurological disorders other than chronic balance disorders, as determined by medical history and neurological screening procedure.
* Any medical condition as determined by the health questionnaire that would interfere with performance on the postural stability evaluation tests.
* Peripheral neuropathies of the lower extremities.
* Subjects who are unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests, and return to clinic for a follow-up visit.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Goebel, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7/10/2009 through 6/30/2012 from Dr. Goebel's clinical practice.
Pre-assignment Details: There was no run-in or washout. All participants received the intervention.
Groups:
- Balcap Group: Balcap group
  Balcap group; balance prosthesis : vibrotactile stimulation
  Patients wore a Balcap device that provided a vibrotactile stimulation that felt like a "buzz" either in front, back, or either side of their head when they swayed a certain distance from their "center".
  They wore the device daily and performed specific personalized exercises as prescribed by a physical therapist. They were tested with and without the balcap during tests of balance and postural stability when they first received the balcap and again six weeks later.
  Each patient wore the balcap device a total of six weeks and then returned the device.
Period: Overall Study
Arm/Group | Balcap Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Balcap Group: Each participant received Balcap Tactile prosthesis
Arm/Group | Balcap Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Dynamic Gait Index (DGI) From Baseline to 6 Weeks.
Description: The DGI is designed to measure a patient's functional balance and postural stability on a scale of 0-3 (3 being normal) for each task. A series of 8 tasks including walking on a level surface, walking while changing speeds, walking with head turns, walking then turning, stepping over obstacles, walking around obstacles, and stairs. For a total scale of 0-24.
Time Frame: 6 weeks
Population: The Dynamic Gait Index (DGI) data were analyzed by way of an linear mixed (LM) model. The DGI response data were treated as the dependent observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Balcap Group: Vibrotactile stimulation exercises with the device over a span of 6 weeks
Arm/Group | Balcap Group
Number analyzed (Participants) | 5
units on a scale | 4.3 (0.040)

ADVERSE EVENTS:
Arm/Group | Balcap Group
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No